CLINICAL TRIAL: NCT04294043
Title: A Phase 1b, Multi-center Study of Intravenous (IV) Gallium Nitrate in Patients With Cystic Fibrosis (CF) Who Are Colonized With Nontuberculous Mycobacteria (NTM) (The ABATE Study)
Brief Title: IV Gallium Study for Patients With Cystic Fibrosis Who Have NTM (ABATE Study)
Acronym: ABATE
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Chris Goss (Other)
Collaborators: Cystic Fibrosis Foundation (Other)
Responsible Party: Sponsor-Investigator, Chris Goss, Professor of Medicine and Pediatrics, University of Washington, Seattle Children's Hospital
Organization: Seattle Children's Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ABATE-IP-18; R01FD006848 (FDA)
Record Dates: First submitted 2020-03-01; First posted 2020-03-03 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Nontuberculous Mycobacterium Infection
Keywords: Cystic Fibrosis; Gallium Nitrate; IV Gallium; Nontuberculous mycobacterium; NTM; Mycobacterium abscessus; mycobacterium avium
MeSH Terms: conditions — Mycobacterium Infections, Nontuberculous; Cystic Fibrosis; Mycobacterium avium-intracellulare Infection | interventions — gallium nitrate; Gallium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Infusion of IV Gallium (Experimental): Gallium nitrate will be infused continuously over 5 days at 200 mg/m2/day. Study drug will be administered via a peripheral IV catheter, a peripherally inserted central catheter (PICC) line, midline catheter, or a chronic indwelling vascular access device using an ambulatory infusion pump infused over 24 hours for 5 sequential days for each cycle. There is a maximum of 2 cycles.
  Interventions: Drug: Gallium nitrate

INTERVENTIONS:
Drug: Gallium nitrate — Study subjects will receive an infusion of gallium nitrate.
  Other Names: Ga; GaN3O9; IV gallium; ganite

SUMMARY:
The purpose of this study is to assess the safety and tolerability of two 5-day infusion cycles of IV gallium in adult patients with CF who are infected with NTM.

Funding Source - FDA Office of Orphan Products Development (OOPD)

DETAILED DESCRIPTION:
This is a prospective, multicenter open-label study in adults with CF who are colonized with M. avium complex and/or M. abscessus complex.

Participants are enrolled into one of the two cohorts:

1. Treatment-Naïve NTM Cohort: participants with persistently positive NTM culture results (either M. avium complex, M. abscessus complex, or both M. avium and M. abscessus) who had never been treated for current NTM species or previous treatment was associated with clearance of NTM.
2. Treatment-Refractory NTM Cohort: participants with persistently positive NTM culture results (either M. avium complex, M. abscessus complex, or both M. avium and M. abscessus) whose treatment failed to respond to 12 months of NTM guideline-based therapy or currently receiving treatment with guideline-based antibiotics for > 12 months.

Subjects will receive two 5-day infusion cycles of IV gallium. The study will evaluate the safety and antimycobacterial effect of two 5-day infusions of IV gallium.

ELIGIBILITY:
Inclusion Criteria for Treatment-Naïve NTM Cohort

1. Written informed consent obtained from participant or participant's legal representative
2. Be willing and able to adhere to the study visit schedule and other protocol requirements
3. All genders ≥ 18 years of age at Visit 1
4. Documentation of a CF diagnosis as evidenced by one or more clinical features consistent with the CF phenotype
5. Documentation of persistently positive NTM culture results that are positive for the same species or sub-species (either M. avium complex, M. abscessus complex, or both M. avium and M. abscessus). Persistently positive cultures are those which meet ONE of the following criteria, after first ignoring any negative culture results that occur within 7 days of a positive culture:

   1. The two most recent NTM culture results from sputum or BAL taken at least 28 days apart are positive.

      OR
   2. At least one NTM culture result in the previous 4 months from sputum or BAL is positive. If there are four or more cultures in the last 12-months at least 3 out of the 4 most recent cultures must be positive for NTM. If there are three or fewer cultures in the past 12 months, then at least 2 of the 3 most recent cultures must be positive for NTM even if some of those cultures are more than 12 months ago.
6. Current NTM species or subspecies has never been treated or previous treatment was associated with clearance of NTM and completed > 2 years prior to Day 1
7. FEV1 ≥ 25 % of predicted value at Screening
8. Able to expectorate sputum
9. Clinically stable with no significant changes in health status within 7 days prior to Day 1
10. Enrolled in the CFF Patient Registry (CFF PR)
11. Willing to discontinue chronic azithromycin use for the duration of the study

Inclusion Criteria for Treatment-Refractory NTM Cohort

1. Written informed consent obtained from participant or participant's legal representative
2. Be willing and able to adhere to the study visit schedule and other protocol requirements
3. All genders ≥ 18 years of age at Visit 1
4. Documentation of a CF diagnosis as evidenced by one or more clinical features consistent with the CF phenotype
5. History of current or prior treatment for NTM pulmonary disease with M. abscessus or M avium (or both M. avium and M. abscessus)

   1. Previously received treatment with guideline-based antibiotics for >12 months without having treatment discontinued for reasons of culture clearance OR
   2. Currently receiving treatment with guideline-based antibiotics for >12 months
6. FEV1 ≥ 25 % of predicted value at Screening
7. Able to expectorate sputum
8. Not hospitalized within 7 days prior to Day 1
9. Enrolled in the CFF Patient Registry (CFF PR)
10. Be willing and able to continue guideline-based antibiotic therapy for M. abscessus or M avium (or both M. avium and M. abscessus) concurrent with IV gallium, if currently on treatment

Exclusion Criteria Treatment-Naïve NTM Cohort

1. Any of the following abnormal lab values at screening:

   * Hemoglobin <10g/dL
   * Platelets <100,000/mm3
   * Absolute neutrophil count < 1500/mm3
   * Aspartate transaminase (AST), alanine transaminase (ALT), gamma-glutamyl transferase (GGT), alkaline phosphatase (ALP), or total bilirubin ≥3 x upper limit of normal
   * Serum creatinine > 2.0 mg/dl and ≥1.5 x upper limit of normal
   * Ionized calcium ≤ lower limit of normal (only performed if total calcium is ≤ lower limit of normal)
2. History of solid organ or hematological transplantation
3. Use of bisphosphonates within 7 days prior to Day 1
4. Known sensitivity to gallium
5. Use of any investigational drug and/or participated in any interventional clinical trial within 28 days prior to Day 1
6. In the opinion of the Investigator, features of active NTM disease are present (e.g., clinical worsening is likely due to NTM disease despite definitive treatment of co-pathogens and/or acute exacerbations)
7. Undergoing treatment for NTM disease or anticipate beginning treatment within 3 months
8. Current diagnosis of osteoporosis
9. For people of childbearing potential:

   * Positive pregnancy test at Visit 1 or
   * Lactating or
   * Unwilling to practice a medically acceptable form of contraception (acceptable forms of contraception: abstinence, hormonal birth control, intrauterine device, or barrier method plus a spermicidal agent), unless surgically sterilized or postmenopausal during the study
10. For people able to father a child: unwilling to use adequate contraception (as determined by the investigator) during the study
11. Has any other condition that, in the opinion of the Site Investigator/designee, would preclude informed consent or assent, make study participation unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving the study objectives
12. New initiation of chronic CF therapy (e.g., CFTR modulators, ibuprofen, azithromycin, inhaled tobramycin, Cayston, etc.) within 28 days prior to Visit 1 (Day 1)
13. Use of azithromycin within 14 days prior to the screening visit

Exclusion Criteria Treatment-Refractory NTM Cohort

1. Any of the following abnormal lab values at screening:

   * Hemoglobin <10g/dL
   * Platelets <100,000/mm3
   * Absolute neutrophil count < 1500/mm3
   * Aspartate transaminase (AST), alanine transaminase (ALT), gamma-glutamyl transferase (GGT), alkaline phosphatase (ALP), or total bilirubin ≥3 x upper limit of normal
   * Serum creatinine > 2.0 mg/dL and ≥1.5 x upper limit of normal
   * Ionized calcium ≤ lower limit of normal (only performed if total calcium is ≤ lower limit of normal)
2. History of solid organ or hematological transplantation
3. Use of bisphosphonates within 7 days prior to Day 1
4. Known sensitivity to gallium
5. Use of any investigational drug and/or participated in any interventional clinical trial within 28 days prior to Day 1
6. Current diagnosis of osteoporosis
7. For people of childbearing potential:

   * Positive pregnancy test at Visit 1 (Day 1) or
   * Lactating or
   * Unwilling to practice a medically acceptable form of contraception (acceptable forms of contraception: abstinence, hormonal birth control, intrauterine device, or barrier method plus a spermicidal agent), unless surgically sterilized or postmenopausal during the study
8. For people able to father a child: unwilling to use adequate contraception (as determined by the investigator) during the study
9. Has any other condition that, in the opinion of the Site Investigator/designee, would preclude informed consent or assent, make study participation unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving the study objectives
10. New initiation of chronic CF therapy (e.g., CFTR modulators, ibuprofen, inhaled tobramycin, Cayston, etc.) within 28 days prior to Visit 1 (Day 1)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-06-17 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Adverse Events of Special Interest | Baseline to Day 57
  Proportion of patients experiencing one or more Adverse Events of Special Interest (AESI). AESIs include the occurrence of either (1) a serious adverse event (SAE) of grade 3 or higher including hospitalizations or (2) study drug discontinuation because of an AE.

SECONDARY OUTCOMES:
Clinically significant abnormal laboratory measures. (safety) | Baseline to Day 57
  Proportion of patients experiencing clinically significant abnormal laboratory measures. Clinically significant abnormal laboratory measures are identified by the site investigator.
NTM clearance (efficacy) | Day 6 to Day 111
  Proportion of subjects who were NTM culture positive at baseline and have at least 2 sequential negative NTM cultures between visits 2 (Day 6) and 7 (Day 111). Those negative cultures must be at least 2 weeks apart.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher H. Goss, MD, MSc, Principal Investigator — University of Washington, Seattle Children's Hospital
Locations (10):
- United States (10):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - National Jewish Health, Denver, Colorado
  - Johns Hopkins University, Baltimore, Maryland
  - The Minnesota Cystic Fibrosis Center, Minneapolis, Minnesota
  - Nationwide Children's Hospital, Columbus, Ohio
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Texas Southwestern, Dallas, Texas
  - University of Vermont Medical Center, Burlington, Vermont
  - University of Washington Medical Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No